CLINICAL TRIAL: NCT01957124
Title: Treatment of the Hypertensive Leg Ulcers by PRF Application
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 5377
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Hypertensive Leg Ulcer
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRF application (Experimental)
  Interventions: Procedure: PRF (Platelet-Rich Fibrin)

INTERVENTIONS:
Procedure: PRF (Platelet-Rich Fibrin)

SUMMARY:
Hypertensive leg ulcers are very painful and difficult to treat ulcers. Their treatment is not well established.

We want to study the efficacy of PRF applications on the pains related to those ulcers.

PRF (Platelet-Rich Fibrin) is an autologous fibrin clot, obtained extemporaneously from patient's blood, without any additive nor complex manipulation. It contains blood platelets and white blood cells, trapped in fibrin during clot formation.

PRF (Platelet-Rich Fibrin) is form immediately after blood punction in a dry tube, that does not contain any anticoagulant. Coagulation naturally occurs within few minutes, and tubes are placed in a centrifuge: red blood cells are separated from the fibrin clot thanks to difference of density, and blood platelets and white blood cells are trapped in the fibrin clot.

The fibrin clot is then rapidly applicated on the ulcer surface for four days. Our hypothesis is that platelet growth factors and cytokines, liberated during platelet activation, could help to treat hypertensive leg ulcers, that are caused by a vascular spasm.

DETAILED DESCRIPTION:
2 to 8 PRF (depending on the ulcer surface), applied on painful hypertensive leg ulcer, and covered by a dressing for 4 days.

Afterwards, dressings are made in a classical way. If needed (persistence of important pain), the PRF application can be repeated after 7 days.

ELIGIBILITY:
Inclusion Criteria:

* hypertensive leg ulcer
* important pain (>= 5/10)

Exclusion Criteria:

* significant venous deficiency
* significant arterial deficiency
* other leg ulcers
* any active diseases such as infection, neoplasia, auto-immune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pain auto evaluation (spontaneous and caused by local care) | Pain was assessed by self-assessment Single Digital Scale - Pain felt in the past 24 hours;
  - Pain experienced during the last ulcer care.
  Ulcers are described using the:
  * Size
  * Presence or absence of necrosis on the bottom and banks
  * Presence or absence of purplish banks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Nicolas Scrivener, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires, Strasbourg, France